CLINICAL TRIAL: NCT05643326
Title: Markers of Clinical and Biological Response to Home Delivered Transcranial Alternating Current Stimulation (tACS) in Patients With Alzheimer's Disease
Brief Title: At Home Gamma tACS in Alzheimer's Disease (tACS@Home)
Acronym: tACS@Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Barbara Borroni, Prof., Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP5395
Record Dates: First submitted 2022-11-24; First posted 2022-12-08 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Real tACS - Real tACS (Experimental): 42 sessions of 40 Hz transcranial alternating current stimulation (5 days/week for 9 weeks) followed by an open-label 42 sessions of 40 Hz transcranial alternating current stimulation (5 days/week for 9 weeks).
  Interventions: Device: 40 Hz transcranial alternating current stimulation
- Sham tACS - Real tACS (Sham Comparator): 42 sessions of sham stimulation (5 days/week for 9 weeks) followed by an open-label 42 sessions of 40 Hz transcranial alternating current stimulation (5 days/week for 9 weeks).
  Interventions: Device: 40 Hz transcranial alternating current stimulation; Device: Sham stimulation

INTERVENTIONS:
Device: 40 Hz transcranial alternating current stimulation — 42 sessions of 40 Hz transcranial alternating current stimulation (5 days/week for 9 weeks)
Device: Sham stimulation — 42 sessions of sham stimulation (5 days/week for 9 weeks)
  Arms: Sham tACS - Real tACS

SUMMARY:
Brain oscillations are ubiquitous in the human brain and have been implicated in cognitive and behavioral states defined in precisely tuned neural networks. In neurodegenerative disorders, neurodegeneration is accompanied by changes in oscillatory activity leading to the emerging concept of neurological and psychiatric disorders as "oscillopathies". Alzheimer's disease, which accounts for the vast majority of age-related dementias, is characterised by a prominent disruption of oscillations in the gamma frequency band. The restoration of gamma oscillations by neural entrainment in animal models of Alzheimer's disease have shown a remarkable decrease in the pathological burden of amyloid and tau via increased microglial activity, resulting in a significant increase of cognitive performances.

Transcranial alternating current brain stimulation (tACS), is a neurophysiological method of non-invasive modulation of the excitability of the central nervous system that is having an increasingly numerous spectrum of potential therapeutic applications. Recent studies have demonstrated the effectiveness of this method in modulating the natural frequencies of cerebral oscillation, underlying multiple cognitive processes such as verbal memory, perception and working memory.

On the basis of these premises, the treatment with gamma tACS is proposed in patients affected by Alzheimer's disease.

In this randomized, double-blind, sham-controlled study, followed by an open-label phase, the investigators will evaluate whether a 9- or 18-weeks treatment with gamma tACS over the precuneus, delivered at home, can improve symptoms in patients with mild Alzheimer's disease.

DETAILED DESCRIPTION:
Brain oscillations are ubiquitous in the human brain and have been implicated in cognitive and behavioral states defined in precisely tuned neural networks. In neurodegenerative disorders, neurodegeneration is accompanied by changes in oscillatory activity leading to the emerging concept of neurological and psychiatric disorders as "oscillopathies". Alzheimer's disease, which accounts for the vast majority of age-related dementias, is characterised by a prominent disruption of oscillations in the gamma frequency band. The restoration of gamma oscillations by neural entrainment in animal models of Alzheimer's disease have shown a remarkable decrease in the pathological burden of amyloid and tau via increased microglial activity, resulting in a significant increase of cognitive performances.

Transcranial alternating current brain stimulation (tACS), is a neurophysiological method of non-invasive modulation of the excitability of the central nervous system that is having an increasingly numerous spectrum of potential therapeutic applications. Recent studies have demonstrated the effectiveness of this method in modulating the natural frequencies of cerebral oscillation, underlying multiple cognitive processes such as verbal memory, perception and working memory.

On the basis of these premises, the treatment with gamma tACS is proposed in patients affected by Alzheimer's disease.

In this randomized, double-blind, sham-controlled study, followed by an open-label phase, the investigators will evaluate whether a 9- or 18-weeks treatment with gamma tACS over the precuneus, delivered at home, can improve symptoms in patients with mild Alzheimer's disease.

Subjects will be randomized in two groups in the first part of the trial. One group will receive a two-months treatment with gamma tACS (40 Hz) over the precuneus while the other group will receive placebo (sham) stimulation. After two-months, both group will undergo real stimulation (open-label phase) with gamma tACS (40 Hz) over the precuneus for two-months. Modulators of response will be considered.

ELIGIBILITY:
Inclusion Criteria for the Patient:

* Mild Alzheimer's disease (CDR 0.5 - 1)

Exclusion Criteria for the Patient:

* Cerebrovascular disorders
* Previous stroke
* Hydrocephalus
* Intra-cranial mass documented by MRI
* History of traumatic brain injury or other neurological diseases
* Serious medical illness other than AD
* History of seizures
* Pregnancy
* Metal implants in the head (except dental fillings)
* Electronic implants (i.e. pace-maker, implanted medical pump)
* Age <18 years

Inclusion Criteria for the Caregiver:

* Age > 18 years
* Compliance in participation in training on the use of the therapeutic device
* Mini-Mental State Examination >26/30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-12-10 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Safety of transcranial alternating current stimulation delivered at home | Through study completion, at week 24
  Incidence of Treatment-Emergent Adverse Events as assessed by the incidence of adverse events graded from 1 (mild) to 5 (fatal).
Tolerability of transcranial alternating current stimulation delivered at home | Through study completion, at week 24
  Tolerability will be evaluated with percentage of compliance (number of delivered stimulations divided by number of programmed stimulations times one-hundred). The primary outcome will be reached if compliance will be >90%.
Changes in Clinical Dementia Rating scale (CDR) sum of boxes | Difference between treatments (real and sham) at week 8
  CDR-SB scores range from 0 to 18, with higher scores indicating worse cognition and daily function.
Changes in Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS-Cog)13 | Difference between treatments (real and sham) at week 8
  ADAS-Cog13 scores range from 0 to 85, with higher scores indicating a greater deficit.
Changes in Face-Name Associative Memory Test (FNAT) scores | Difference between treatments (real and sham) at week 8
  The Face-Name Associative Memory Test is a cross-modal associative memory test, it includes 20 face-name pairs. The administration procedure starts with the presentation of 20 faces with each name and participants should read the name underneath the faces and try to learn each face-name pair. After 5 minutes, the faces are shown one by one and participants are asked to recall the associated names from 4 different names. The correct number of pairs recalled is recorded. The score ranges from 0 (worse performance) to 20 (best performance).
Changes in Alzheimer's Disease Assessment Scale Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) | Difference between treatments (real and sham) at week 8
  ADCS-ADL scores range from 0 to 78, with lower scores indicating greater functional impairment.

SECONDARY OUTCOMES:
Changes in Clinical Dementia Rating scale (CDR) sum of boxes | Change from baseline to week 8 - 16 - 24
  CDR-SB scores range from 0 to 18, with higher scores indicating worse cognition and daily function.
Changes in Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS-Cog)13 | Change from baseline to week 8 - 16 - 24
  ADAS-Cog13 scores range from 0 to 85, with higher scores indicating a greater deficit.
Changes in Rey Auditory Verbal Learning Test scores | Change from baseline to week 8 - 16 - 24
  Participants are given a list of 15 unrelated words repeated over five different trials and are asked to repeat. Another list of 15 unrelated words are given and the patient must again repeat the original list of 15 words and then again after 30 minutes. The score ranges from 0 (worse performance) to 15 (best performance).
Changes in Face-Name Associative Memory Test (FNAT) scores | Change from baseline to week 8 - 16 - 24
  The Face-Name Associative Memory Test is a cross-modal associative memory test, it includes 20 face-name pairs. The administration procedure starts with the presentation of 20 faces with each name and participants should read the name underneath the faces and try to learn each face-name pair. After 5 minutes, the faces are shown one by one and participants are asked to recall the associated names from 4 different names. The correct number of pairs recalled is recorded. The score ranges from 0 (worse performance) to 20 (best performance).
Changes in the Neuropsychiatric Inventory (NPI-Q) | Change from baseline to week 8 - 16 - 24
  The NPI-Q is designed to be an informant-based interview that assesses neuropsychiatric symptoms of the participant over the previous month. The score ranges from 0 (no symptoms) to 180 (severe symptoms).
Changes in Caregiver Burden Inventory (CBI) | Change from baseline to week 8 - 16 - 24
  The Caregiver Burden Inventory (CBI) includes 24 items and 5 dimensions: Time-dependence, developmental, physical, emotional, and social burden. There are 5 items for each dimension, except for the physical dimension, which has four items. Each item signifies a score between zero (not descriptive) and four (highly descriptive), with a higher score indicating greater care burden. Therefore the total score for time-dependence, developmental, emotional, and social burden range from 0 to 20 except for physical burden where scores range from 0 to 16. The total score ranges from 0 (no burden) to 96 (severe burden).
Changes in Alzheimer's Disease Assessment Scale Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) | Change from baseline to week 8 - 16 - 24
  ADCS-ADL scores range from 0 to 78, with lower scores indicating greater functional impairment.
Change in SAI measurements | Change from baseline to week 8 - 16 - 24
  By using transcranial magnetic stimulation (TMS), the investigators will evaluate the effects of gamma tACS on short latency afferent inhibition (SAI), which is a marker of cholinergic transmission. SAI is expressed as % of the unconditioned motor evoked potential.
Change in EEG gamma power | Change from baseline to week 8 - 16 - 24
  By using electroencephalography (EEG), the investigators will evaluate the change in gamma power.
Change in plasma NfL levels | Change from baseline to week 8 - 16 - 24
  Changes in plasma neurofilament light (NfL) levels (pg/mL) will be evaluated.
Change in plasma GFAP levels | Change from baseline to week 8 - 16 - 24
  Changes in plasma glial fibrillary acidic protein (GFAP) levels (pg/mL) will be evaluated.
Change in plasma amyloid beta1-40 levels | Change from baseline to week 8 - 16 - 24
  Change in plasma amyloid beta1-40 levels (pg/mL) will be evaluated.
Change in plasma amyloid beta1-42 levels | Change from baseline to week 8 - 16 - 24
  Change in plasma amyloid beta1-42 levels (pg/mL) will be evaluated.
Change in plasma pTau217 | Change from baseline to week 8 - 16 - 24
  Change in plasma pTau217 levels (pg/mL) will be evaluated.
Change in resting state MRI connectivity | Change from baseline to week 8
  Change in resting state magnetic resonance imaging connectivity (default mode network) both static and dynamic.
Change in plasma TMT part B scores | Change from baseline to week 8 - 16 - 24
  The Trail Making Test Part B consists of 24 circles on a piece of paper, but rather than all of the circles containing numbers, half of the circles have the numbers 1-12 in them and the other half (12) contain the letters A-L. The person taking the test has to draw a line from one circle to the next in ascending order; however, he must alternate the circles with numbers in them (1-13) with circles with letters in them (A-L). In other words, he is to connect the circles in order like this: 1-A-2-B-3-C-4-D-5-E and so on. Scoring is based on time taken to complete the test with lower scores being better.
Changes in semantic fluency task | Change from baseline to week 8 - 16 - 24
  In the semantic fluency task, participants are asked to generate as many words as possible from a given category (animals) within a limited time (60 seconds); lower scores indicate greater impairment in verbal fluency.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Borroni, MD, Principal Investigator — Azienda Ospedaliera Spedali Civili, Brescia; Alberto Benussi, MD, Principal Investigator — University or Brescia
Locations (1):
- ASST Spedali Civili di Brescia, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fries P. Neuronal gamma-band synchronization as a fundamental process in cortical computation. Annu Rev Neurosci. 2009;32:209-24. doi: 10.1146/annurev.neuro.051508.135603. PMID 19400723
- [Background] Iaccarino HF, Singer AC, Martorell AJ, Rudenko A, Gao F, Gillingham TZ, Mathys H, Seo J, Kritskiy O, Abdurrob F, Adaikkan C, Canter RG, Rueda R, Brown EN, Boyden ES, Tsai LH. Gamma frequency entrainment attenuates amyloid load and modifies microglia. Nature. 2016 Dec 7;540(7632):230-235. doi: 10.1038/nature20587. PMID 27929004
- [Background] Adaikkan C, Middleton SJ, Marco A, Pao PC, Mathys H, Kim DN, Gao F, Young JZ, Suk HJ, Boyden ES, McHugh TJ, Tsai LH. Gamma Entrainment Binds Higher-Order Brain Regions and Offers Neuroprotection. Neuron. 2019 Jun 5;102(5):929-943.e8. doi: 10.1016/j.neuron.2019.04.011. Epub 2019 May 7. PMID 31076275
- [Background] Martorell AJ, Paulson AL, Suk HJ, Abdurrob F, Drummond GT, Guan W, Young JZ, Kim DN, Kritskiy O, Barker SJ, Mangena V, Prince SM, Brown EN, Chung K, Boyden ES, Singer AC, Tsai LH. Multi-sensory Gamma Stimulation Ameliorates Alzheimer's-Associated Pathology and Improves Cognition. Cell. 2019 Apr 4;177(2):256-271.e22. doi: 10.1016/j.cell.2019.02.014. Epub 2019 Mar 14. PMID 30879788
- [Background] Herrmann CS, Rach S, Neuling T, Struber D. Transcranial alternating current stimulation: a review of the underlying mechanisms and modulation of cognitive processes. Front Hum Neurosci. 2013 Jun 14;7:279. doi: 10.3389/fnhum.2013.00279. eCollection 2013. PMID 23785325
- [Background] Benussi A, Cantoni V, Cotelli MS, Cotelli M, Brattini C, Datta A, Thomas C, Santarnecchi E, Pascual-Leone A, Borroni B. Exposure to gamma tACS in Alzheimer's disease: A randomized, double-blind, sham-controlled, crossover, pilot study. Brain Stimul. 2021 May-Jun;14(3):531-540. doi: 10.1016/j.brs.2021.03.007. Epub 2021 Mar 21. PMID 33762220
- [Background] Benussi A, Cantoni V, Grassi M, Brechet L, Michel CM, Datta A, Thomas C, Gazzina S, Cotelli MS, Bianchi M, Premi E, Gadola Y, Cotelli M, Pengo M, Perrone F, Scolaro M, Archetti S, Solje E, Padovani A, Pascual-Leone A, Borroni B. Increasing Brain Gamma Activity Improves Episodic Memory and Restores Cholinergic Dysfunction in Alzheimer's Disease. Ann Neurol. 2022 Aug;92(2):322-334. doi: 10.1002/ana.26411. Epub 2022 Jun 6. PMID 35607946
- [Derived] Cantoni V, Casula EP, Tarantino B, Cupidi C, Huber N, Altomare D, Premi E, Zummo E, Esposito R, Leonardi C, Herukka SK, Solje E, Ferrari A, Cotelli MS, Gasparotti R, Martorana A, Fracassi C, Santarnecchi E, Koch G, Haapasalo A, Grassi M, Benussi A, Borroni B. Home-Based Gamma Transcranial Alternating Current Stimulation in Patients With Alzheimer Disease: A Randomized Clinical Trial. JAMA Netw Open. 2025 Dec 1;8(12):e2546556. doi: 10.1001/jamanetworkopen.2025.46556. PMID 41359335